CLINICAL TRIAL: NCT01150500
Title: RESOLUTE JAPAN SVS: The Clinical Evaluation of the MDT-4107 Drug-Eluting Coronary Stent in the Treatment of De Novo Lesions in Small Diameter Native Coronary Arteries
Brief Title: RESOLUTE Japan SVS: The Clinical Evaluation of the MDT-4107 DES in the Treatment of De Novo Lesions in Small Diameter Native Coronary Arteries
Acronym: RJ-SVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT2-07-05
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Arterial Occlusive Diseases; Myocardial Ischemia; Cardiovascular Diseases; Coronary Artery Disease
Keywords: Medtronic; Japan; Arterial Occlusive Diseases; Myocardial Ischemia; Cardiovascular Diseases; Coronary Artery Disease; Small Vessel Stent
MeSH Terms: conditions — Arterial Occlusive Diseases; Myocardial Ischemia; Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Eluting Stent (Experimental): Up to two lesions in two separate target vessels may be treated under this protocol. The lesions should be amenable to treatment with at least one 2.25 mm stent, a second lesion could be treated with any stent from 2.25 to 3.5 mm.
  Interventions: Device: MDT-4107 Zotarolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: MDT-4107 Zotarolimus-Eluting Coronary Stent
  Other Names: Endeavor Resolute, Zotarolimus Drug Eluting Stent, Medtronic

SUMMARY:
The objective of the study is To verify the safety and efficacy of the MDT-4107 Drug-Eluting Coronary Stent in the treatment of de novo lesions in native coronary arteries with a reference vessel diameter (RVD) that allows the use of 2.25mm diameter stents.

DETAILED DESCRIPTION:
The objective of the study is to verify the safety and efficacy of the MDT-4107 Drug-Eluting Coronary Stent in the treatment of de novo lesions in native coronary arteries with a reference vessel diameter (RVD) that allows the use of 2.25mm diameter stents.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable candidate for percutaneous coronary intervention (PCI),stenting, and emergency coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia and/or positive functional study
* Informed consent
* Patient agrees to comply with specified follow-up evaluations at same investigational site
* Single target lesion or two target lesions located in separate coronary arteries
* De novo lesion(s) in native coronary artery(ies)
* Target lesion(s) ≤ 27 mm in length
* Target vessel(s) have reference vessel diameter 2.25 mm to 3.5 mm

Exclusion Criteria:

* Within 7 days of implant platelet count <100,000 cells/mm³ or >700,000 cells/mm³; White Blood Cell (wbc) count <3,000 cells/mm³; serum creatinine level >2.5 mg/dl
* Acute myocardial infarction (MI) within 72 hrs of the index procedure (Q wave myocardial infarction(QWMI)/non Q wave myocardial infarction (NQMI) or any elevation of creatinine kinease myocardial-band isoenzyme(CK-MB) > lab upper limit of normal)
* Previous PCI of target vessel(s) within 9 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of target vessel(s) within 12 months post-index procedure
* History of stroke or transient ischemic attack(TIA) within prior 6 months
* Participating in investigational drug/device study that has not completed primary endpoint or interferes with study endpoints
* Inability to comply with required trial antiplatelet regimen
* Previous stent in target vessel unless it has been at least 9 months since stent placed and target lesion(s) is/are at least 15 mm from previous stent
* Target vessel(s) has/have other lesions w/ > 40% diameter stenosis
* Unprotected left main coronary artery disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Sohana Kamakura General Hosptial
Locations (1):
- Shonan Kamakura General Hospital, Kanagawa, Japan

REFERENCES:
- [Derived] Saito S, Maehara A, Vlachojannis GJ, Parise H, Mehran R; RESOLUTE Japan Investigators. Clinical and angiographic evaluation of the resolute zotarolimus-eluting coronary stent in Japanese patients - long-term outcome in the RESOLUTE Japan and RESOLUTE Japan small vessel study. Circ J. 2015;79(1):96-103. doi: 10.1253/circj.CJ-14-0836. Epub 2014 Nov 27. PMID 25428602
- See also: Medtronic Clinical Trials Link — http://clinicaltrials.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study the first patient was enrolled in June 2011 and the last patient was enrolled in January 2012 in eleven hospitals in Japan.
Pre-assignment Details: There was no significant episode for screening processes.
Groups:
- Stent Placement: Up to two lesions in two separate target vessels may be treated under this protocol. The lesions should be amenable to treatment with at least one 2.25 mm stent, a second lesion could be treated with any stent from 2.25 to 3.5 mm.
  MDT-4107 Zotarolimus-Eluting Coronary Stent : Implantation of a MDT-4107 Zotarolimus-Eluting Coronary Stent
Period: Overall Study
Arm/Group | Stent Placement
Started | 65
Completed | 0
Not Completed | 65

BASELINE CHARACTERISTICS:
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 44
Region of Enrollment [Number; unit: participants]
  Japan | 65

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure(TLF)
Description: Target Lesion Failure (TLF) at 9 months post-procedure defined as a composite measure of cardiac death, heart attack attributed to the target vessel (target vessel myocardial infarction), and ischemia-driven target lesion revascularization (TLR)
Time Frame: 9 month
Population: All 65 patients enrolled were analyzed as intent-to-treat (ITT) population and per protocol(PP) population.
Measure: Number; unit: percentage of TLF
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
percentage of TLF | 4.62

2. Secondary Outcome: MACE (Major Adverse Cardiac Event)
Description: Death, myocardial infarction (Q-wave and non-Q-wave), emergent coronary bypass, or clinically-driven repeat target lesion revascularization by percutaneous surgical methods.
Time Frame: Baseline and 9 month
Population: 65 patients were analyzed as ITT population
Measure: Number; unit: percentage of patient
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
percentage of patient | 2

3. Secondary Outcome: Late Lumen Loss
Description: Defined as the difference between the post-procedure immediate minimal lumen diameter (MLD) and the follow-up angiography MLD at 9 month.
Time Frame: Baseline and 9 months
Population: 67 Lesions in 65 patients are analysed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
mm | 0.27 (0.33)

4. Secondary Outcome: Binary Angiographic Restenosis
Description: Defined as => 50% in-stent diameter stenosis at the follow-up angiogram at 9 month. If an in-stent measurement is not available, the in-lesion diameter was used.
Time Frame: Baseline and 9 month
Population: 67 lesions in 65 patients were analysed.
Measure: Number; unit: percentage of patient
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
percentage of patient | 1.5

5. Secondary Outcome: Minimum Luminal Diameter
Description: The average of two orthogonal views(when possible) of narrowest point within the area of assessment-in lesion, in stent or in segment. minimal luminal diameter is visually estimated during angiography by the investigator; it is measured during quantitative coronary angiography by the Angiographic Core Laboratory.
Time Frame: 9 month
Population: 67 lesions in 65 patient were analyzed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
mm | 1.86 (0.39)

6. Secondary Outcome: Percent Diameter Stenosis
Description: The value calculated as 100 x (Reference Vessel Diameter(RVD) - Minimum luminal diameter(MLD))/ RVD using the mean values from orthogonal views (when possible) by quantitative coronary angiography(QCA).
Time Frame: Baseline and 9 month
Population: 67 lesions in 65 patients were analyzed.
Measure: Mean (Standard Deviation); unit: % DS (diameter stenosis)
Arm/Group | Stent Placement
Number analyzed (Participants) | 65
% DS (diameter stenosis) | 12.92 (14.63)

7. Secondary Outcome: Clinical Endpoints
Description: Success (device, lesion, procedure), major adverse cardiac events (MACE), target vessel failure (TVF), and stent thrombosis
Time Frame: 5 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event (AE) is collected for time between the index procedure and 9 months follow-up.Any serious adverse event (SAE) occurring from the index procedure to 5 year follow-up assessment, regardless of cause, is collected.
Description: Major Cardiac Adverse Event (secondary endpoint) is considered " serious " in this study
Arm/Group | Stent Placement
Serious Adverse Events (participants affected / at risk) | 16/65
Other Adverse Events (participants affected / at risk) | 25/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stent Placement (N=65)
ANGINA PECTORIS (Cardiac disorders) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1)
CATARCT (Eye disorders) | 1 (1)
GASTRIC ULCER HAEMORRAGE (Gastrointestinal disorders) | 1 (1)
MALTI-ORGAN FAILURE (General disorders) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
LUMBER SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1)
ACTIVITY OF DIALY LIVING IMPAIRED (Social circumstances) | 1 (1)
ATERIOSCLEROSIS OBLITERANS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stent Placement (N=65)
NASOPHARYNGITIS (Infections and infestations) | 9 (9)
ANGINA PECTORIS (Cardiac disorders) | 4 (4)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4)
BLOOD TRIGYCERIES INCREASED (Investigations) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No